CLINICAL TRIAL: NCT03238274
Title: Sofia 2 Lyme FIA Whole Blood Clinical Study
Status: Completed | Type: Observational
Sponsor: Quidel Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: CS-0267-01
Record Dates: First submitted 2017-08-01; First posted 2017-08-03 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Borrelia; Infection, Burgdorferi (Erythema Chronicum Migrans)
MeSH Terms: conditions — Glossitis, Benign Migratory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (3):
- Arm 1: Arm 1 is a multi-site, single visit, prospective clinical study where subjects will be enrolled based on a physician's assessment of current Lyme specific symptoms from recent contact with a tick.
  Interventions: Device: Sofia 2 Lyme FIA testing
- Arm 2: Arm 2 will consist of subjects selected from a pool of patients that were previously determined to have Lyme disease either by the presence of the diagnostic rash (erythema migrans) or through laboratory findings and physician diagnosis based on patient symptoms. In this Arm the site may recruit by contacting subjects previously diagnosed with Lyme disease no longer than 16 months post diagnosis and no earlier than 1 week post diagnosis.
  Interventions: Device: Sofia 2 Lyme FIA testing
- Arm 3: Arm 3 will consist of subjects selected from a pool of patients that were previously determined to have Lyme disease either by the presence of the diagnostic rash (erythema migrans) or through laboratory findings and physician diagnosis based on patient symptoms. In this Arm the site may recruit by contacting subjects previously diagnosed with Lyme disease between 17 months and 50 months post diagnosis. For the subject to be enrolled, a physician must have diagnosed the subject to have Lyme disease based on clinical symptoms.
  Interventions: Device: Sofia 2 Lyme FIA testing

INTERVENTIONS:
Device: Sofia 2 Lyme FIA testing — IVD testing of whole blood or serum/plasma to aid in the detection of anti-B. burgdorferi IgG / IgM antibody

SUMMARY:
The objective of this study is to demonstrate the clinical performance of the Sofia® 2 analyzer and Sofia Lyme FIA test in the CLIA waived test environment in comparison to Comparator Method(s) and/or an FDA cleared predicate test(s) using matched finger-stick, whole blood and serum from symptomatic subjects.

DETAILED DESCRIPTION:
The objective of this study is to demonstrate the clinical performance of the Sofia® 2 analyzer and Sofia Lyme FIA test in the CLIA waived test environment in comparison to Comparator Method(s) and/or an FDA cleared predicate test(s) using matched finger-stick, whole blood and serum from symptomatic subjects. The finger-stick and venous whole blood specimens will be tested by CLIA waived test operators. The matched plasma (from the leftover whole blood) and serum specimens will be sent to a separate reference laboratory for testing to compare the matched specimen using the Comparator Method(s) and/or an FDA-cleared predicate test(s). The results of this study may be used to support a 510(k) and/or CLIA-Waiver submission for testing whole blood sample types.

ELIGIBILITY:
Inclusion Criteria:

* Arm 1 - Prospective symptomatic subjects, must have had a known or suspected exposure or tick-bite from an endemic area prior to onset of symptoms, and be currently exhibiting the following:
* The physician determines that the subject has an expanding erythema migrans (EM) lesion or "bulls-eye rash" with evidence of clearing in the center and has requested 2 tier serological testing or prescribed a ≥10 day course of antibiotics such as doxycycline in subjects > 8 years old or amoxicillin, cefuroxime or doxycycline in subjects ≤8 years of age:

Or

- The physician must observe current symptoms, including:

At least three (3) of the listed acute stage symptoms listed:

* fatigue
* night sweats
* chills
* fever
* headache
* arthralgia
* mildly stiff neck
* myalgia i. one or more symptoms a. through h. are determined to be intermittent

Or,

* at least one (1) of the following current conditions:
* recurrent, brief attacks (weeks/months) of objective joint swelling in one or more joints, sometimes followed by chronic arthritis in one or a few joints,
* lymphocytic meningitis
* cranial neuritis (partial facial palsy and may be bilateral)
* radiculoneuropathy
* encephalomyelitis
* acute onset of high-grade (2nd or 3rd degree) atrioventricular conduction defects that resolve in days to weeks, sometimes associated with myocarditis

In addition, the physician must be sufficiently confident in the possibility of Lyme disease to have requested two-tier diagnostic testing and/or prescribed a ≥10 day course of antibiotics such as doxycycline in patients > 8 years old or amoxicillin, cefuroxime or doxycycline in patients ≤8 years of age.

Arm 2 - Previously diagnosed with Lyme disease / confirmed case of Lyme disease: Within the past 16 months, a physician must have previously diagnosed the subject based on the presence of an EM rash or based on symptoms and confirmed by laboratory findings as outlined in the CDC two Tier Testing algorithm. A copy of the subject's medical record documenting the diagnosis must be obtained, and kept as source documentation at the enrolling site.

Arm 3 - Previously diagnosed with Lyme disease / confirmed case of Lyme disease: Within the past 17 to 50 months, a physician must have previously diagnosed the subject based on the presence of an EM rash or based on symptoms and confirmed by laboratory findings as outlined in the CDC two Tier Testing algorithm. A copy of the subject's medical record documenting the diagnosis must be obtained, and kept as source documentation at the enrolling site.

Exclusion Criteria:

* Unable to understand and consent to participation; for minors this includes parent or legal guardian.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Known or suspected exposure or tick-bite from an endemic area prior to onset of symptoms
Sampling Method: Probability Sample
Enrollment: 597 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Detection of anti-B. burgdorferi IgG / IgM antibody | 15 minutes
  Accurate detection of presence or absence of anti-B. burgdorferi IgG / IgM antibody

CONTACTS AND LOCATIONS:
Overall Officials: Tom Clement, Study Director — Quidel Corporation
Locations (11):
- United States (11):
  - NECCR Primacare Research, LLC, Fall River, Massachusetts
  - Main Road Family Medicine, South Westport, Massachusetts
  - Essentia Institute of Rural Health, Duluth, Minnesota
  - Regional Clinical Research, Endwell, New York
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Harleysville Medical Associates, Harleysville, Pennsylvania
  - Lincoln Primary Care, Lincoln, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island
  - Center for Medical Research, LLC, Providence, Rhode Island
  - Ocean State Primary Care, Westerly, Rhode Island
  - Marshfield Clinic Research Institute, Marshfield, Wisconsin

IPD SHARING:
Plan to Share IPD: No
There is no plan or intention to share participant data with others.